CLINICAL TRIAL: NCT01884675
Title: A Randomised, Multicentre, Double-Blind, Placebo-Controlled Study Of Ambrisentan In Subjects With Inoperable Chronic Thromboembolic Pulmonary Hypertension (CTEPH).
Brief Title: Ambrisentan for Inoperable Chronic Thromboembolic Pulmonary Hypertension.
Acronym: AMBER I
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115811
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Endothelin Receptor Antagonist; Inoperable Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Hypertension | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambrisentan (Experimental): Subjects in this arm will receive ambrisentan 5 mg tablet once daily during the treatment period.
  Interventions: Drug: Ambrisentan 5 mg
- Placebo (Placebo Comparator): Subjects in this arm will receive ambrisentan-matching placebo tablet once daily during the treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan 5 mg — White, film-coated, immediate-release tablets, containing 5 mg ambrisentan for single dose oral.
  Arms: Ambrisentan
Drug: Placebo — White, film-coated, ambrisentan-matching placebo tablet for single oral dose
  Arms: Placebo

SUMMARY:
It is hypothesised that ambrisentan may provide benefit to subjects with inoperable chronic thromboembolic pulmonary hypertension (CTEPH), where currently no proven or licensed treatment options exist. This Phase III, randomized, double-blind placebo controlled parallel group, 16 week study will compare the safety and efficacy of ambrisentan 5 milligrams (mg) versus placebo in subjects with inoperable CTEPH. The study will enrol 160 subjects, to assure at least 72 evaluable subjects per treatment arm, based on 10% drop-out rate.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to beginning study-related procedures.
* Subject must be between 18-80 years of age, inclusive, at the Screening Visit.
* Subjects must have a diagnosis of CTEPH at an expert centre with a positive V/Q and CT angiogram and a pulmonary angiogram if available within 6 months prior to screening.
* Subject must meet all of the following haemodynamic criteria by means of a RHC within 3 months prior to screening: Mean pulmonary artery pressure (mPAP) of >25 millimeters of mercury (mmHg), Pulmonary vascular resistance (PVR) >400 dynes.sec/centimetre (cm)^5, Pulmonary capillary wedge pressure (PCWP) or Left ventricle end diastolic pressure (LVEDP) of <15 mmHg.
* Subjects must have previously been judged inoperable due to the obstruction being surgically inaccessible (i.e. distal disease) by an expert multidisciplinary team which must include at least one cardiology or respiratory consultant, and one consultant PEA surgeon. For countries with CTEPH expert centers [including at least a surgeon with sound experience performing Pulmonary Endarterectomy (PEAs)] the expert team will be the local expert centre. For countries without a CTEPH surgical expert center a central adjudication committee will assess the operability of the subjects during the screening period.
* Subject must walk a distance of >150 Meters (m) and < 475 m at the screening visit.
* Subject must have a current diagnosis of being in WHO Functional Class II or III.
* Subject, with or without supplemental oxygen, must have a resting arterial oxygen saturation (SaO2) > 92% as measured by pulse oximetry at the Screening Visit.
* Subjects must have received anticoagulation for a minimum of 3 months prior to Screening
* Female subject of childbearing potential must agree to use 2 reliable methods of contraception from the Screening Visit until study completion and for at least 30 days following the last dose of Investigational Product
* Subject must agree not to participate in a clinical study involving another investigational drug or device throughout this study.
* Subject must be competent to understand the information given in the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved informed consent form (ICF) and must sign the form prior to the initiation of any study procedures.

Exclusion Criteria:

* Subject received previous Pulmonary arterial hypertension (PAH) therapy (Phosphodiesterase type 5 [PDE5i], Endothelin receptor antagonist [ERA], chronic prostanoid use)
* Subject has previously discontinued other ERA in either another clinical study or commercial product for safety or tolerability reasons other than for liver function abnormalities.
* Subject has a known hypersensitivity to the Investigational Products, the metabolites, or formulation excipients
* Subject has previously undergone a pulmonary endarterectomy or a balloon pulmonary angioplasty
* Subject receiving intravenous inotropes within 2 weeks prior to the Screening Visit (e.g. dopamine, dobutamine)
* Subjects receiving Calcium Channel Blockers or 5-hydroxy-3-methylglutaryl-coenzyme A 5-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors (i.e., statins) on an unstable dose 4 weeks prior to the Screening Visit (to be eligible subjects must not have changed their dose <4 weeks prior to the screening visit)
* Subject has not enrolled in an exercise training program for cardiopulmonary rehabilitation within 12 weeks prior to the Screening Visit and must agree not to enroll in an exercise training program for pulmonary rehabilitation during the Screening Period and the first 16 weeks of the study. Subjects enrolled in an exercise program for pulmonary rehabilitation 12 weeks prior to screening may enter the study if they agree to maintain their current level of rehabilitation for the first 16 weeks of the study.
* Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) > 3x Upper limit of normal (ULN)
* Bilirubin > 1.5xULN (>35% direct bilirubin)
* Subject has severe renal impairment [estimated creatinine clearance <30 millilitre/minute (mL/min)] at the Screening Visit
* Subject has moderate - severe hepatic impairment (Child-Pugh class B-C with or without cirrhosis) at the Screening Visit
* Subject has clinically significant anaemia: Hemoglobin (Hb) < 10 grams/decilitre (g/dL)
* Subjects with bleeding disorders or significant active peptic ulceration in the opinion of the investigator
* Subject has uncontrolled hypertension (>180/110 mmHg) at screening
* Subject has severe hypotension (<90/50 mmHg) at screening
* Subject has had an acute myocardial infarction within the last 90 days prior to screening
* Subject has, in the opinion of the investigator, clinically significant aortic or mitral valve disease; pericardial constriction; restrictive or congestive cardiomyopathy; life-threatening cardiac arrhythmias; significant left ventricular dysfunction (ejection fraction <50% of normal); left ventricular outflow obstruction; symptomatic coronary artery disease; autonomic hypotension; fluid depletion.
* Subject with significant pulmonary disease Forced expiratory volume in 1 second (FEV1) <70% of predicted): Chronic obstructive pulmonary disease (COPD), Emphysema, evidence of fibrotic lung disease on imaging
* Subject has clinically significant fluid retention in the opinion of the investigator
* Subject with significant obesity [Body mass index (BMI) ≥35], cardiovascular, musculoskeletal or any other condition that in the opinion of the investigator may involve an impairment of exercise capacity or the performance of the 6MWD test (e.g. previous history of hip/knee surgery, lower limb ulcers associated with autoimmune diseases)
* Subject with cardiovascular, liver, renal, haematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease that, in the opinion of the Investigator, may adversely affect the safety of the subject and/or efficacy of the investigational product or severely limit the lifespan of the subject other than the condition being studied
* Subjects with a prior malignancy whose cancer is expected to require additional active treatment in the next 2 years and whose prior malignancy would prevent them from fully participating in the study
* Female subject who is pregnant or breastfeeding
* Subject has demonstrated noncompliance with previous medical regimens
* Subject has a recent (within 1 year) history of abusing alcohol or illicit drugs
* Subject has participated in a clinical study involving another investigational drug or device within 4 weeks before the Screening Visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (2):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Dallas, Texas
- Argentina (4):
  - GSK Investigational Site, Corrientes, Corrientes Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santa Fe, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Austria (3):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, London, Ontario
- China (4):
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
- GSK Investigational Site, Prague, Czechia
- Germany (7):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
- Israel (2):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Zrifin
- Japan (7):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Monterrey NL, Nuevo León, Mexico
- GSK Investigational Site, Amsterdam, Netherlands
- Russia (3):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Tomsk
- GSK Investigational Site, Riyadh, Saudi Arabia
- GSK Investigational Site, Seoul, South Korea
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Seville
- United Kingdom (3):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Clydebank
  - GSK Investigational Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 160 participants were planned to be enrolled, however only 33 participants were randomized in the study.
Pre-assignment Details: This was a double-blind study which included clinic visits at Screening, Baseline visit, Weeks 4, 8, 12 and 16. A Follow-up visit was scheduled approximately 30 days after the Week 16 visit for those participants not continuing into study AMB116457 (Open-label extension study).
Groups:
- Placebo: Participants received a matching placebo tablet once daily for a period of 16 weeks.
- Ambrisentan 5mg: Participants received an ambrisentan 5milligram (mg) tablet, once daily for a period of 16 weeks.
Period: Overall Study
Arm/Group | Placebo | Ambrisentan 5mg
Started | 16 | 17
Completed | 13 | 15
Not Completed | 3 | 2
Not completed — Study closed/terminated | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ambrisentan 5mg | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 59.0 (8.99) [51.0 to 66.5] | 63.0 (13.38) [51.0 to 71.0] | 62.0 (11.31) [51.0 to 68.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 6 | 9 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 6 | 5 | 11
  Asian - Japanese Heritage | 4 | 1 | 5
  White - White/Caucasian/European Heritage | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Six Minutes Walking Distance (6MWD) at Week 16
Description: The 6-minute walk test was conducted according to the American Thoracic Society guidelines in accordance with local standard operating procedures. 6MWD was measured by a 6-minute walk test. This test measures the distance that a participant can walk in a period of 6 minutes. Change from baseline was calculated at Weeks 4, 8, 12 and 16. Change from Baseline was calculated as value at the specified visit minus the Baseline value. Data at Baseline is based on average of two consecutive test results during Screening/Baseline period that differ by <10%. If only one measurement was available, that measurement was used. In any cases where the protocol-defined criteria for Baseline 6MWD was not met, the Baseline value was based on the last two consecutive measurements for a participant.
Time Frame: Baseline (Week 0); Weeks 4, 8, 12 and 16/Early Withdrawal
Population: Intent-to-Treat (ITT) Population: comprised of all randomized participants who received at least 1 dose of study drug. Only those participants with available data at Baseline and the specified timepoint (represented as n=X, X for placebo and ambrisentan respectively) were summarized.
Measure: Median (Inter-Quartile Range); unit: Meters
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Meters
  Week 4, n=15, 17 | 5.00 [-1.50 to 16.50] | 14.00 [1.00 to 42.50]
  Week 8, n=14, 16 | 7.50 [-14.50 to 22.50] | 26.25 [3.25 to 61.25]
  Week 12, n=13, 15 | 5.50 [-23.00 to 39.50] | 20.50 [4.00 to 68.00]
  Week 16, n=13, 15 | -10.00 [-32.50 to 20.00] | 25.00 [12.00 to 49.00]
  Early Withdrawal, n=3, 2 | 7.50 [-46.50 to 43.50] | 41.25 [0.00 to 82.50]

2. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week 16
Description: PVR is a measure of cardiopulmonary haemodynamics. Change from Baseline was calculated as value at specified visit minus Baseline value. Baseline is the last value recorded on or prior to start of study treatment.
Time Frame: Baseline (Week 0) and Week 16
Population: ITT Population. Only those participants with available data at Baseline and the specified timepoint were analysed.
Measure: Median (Inter-Quartile Range); unit: Dynes*second/centimeter^5
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 11 | 13
Dynes*second/centimeter^5 | -103.0 [-122.0 to -88.0] | -130.0 [-502.0 to -78.0]

3. Secondary Outcome: Change From Baseline in WHO Functional Class (FC) at Weeks 4, 8, 12 and 16/Early Withdrawal
Description: The WHO FC indicates the severity of PAH and is an adaptation of the New York Heart Association classification. It was assessed by the investigator. There are four grades for WHO FC based on severity of symptoms (Class I = none, Class IV = most severe). This functional classification system links symptoms with activity limitations, and allows clinicians to quickly predict disease progression and prognosis, as well as the need for specific treatment regimens, irrespective of the underlying etiology of PAH. Baseline is the last value recorded on or prior to start of study treatment. Change from Baseline was calculated as the value at specified visit minus the Baseline value. For analyse purposes, the WHO FC Class categories of I-IV were mapped to a numeric scale of 1-4.
Time Frame: Baseline (Week 0); Weeks 4, 8, 12 and 16/Early Withdrawal
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Groups:
- Ambrisentan 5mg: Subjects in this arm will receive ambrisentan-matching placebo tablet once daily during the treatment period.
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Scores on a scale
  Week 4, n=15, 17 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Week 8, n=14, 16 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Week 12, n=13, 15 | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Week 16, n=13, 15 | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Early Withdrawal, n=3, 2 | 0.0 [-1.0 to 0.0] | 0.0 [0.0 to 0.0]

4. Secondary Outcome: Change From Baseline in Borg CR10 Scale (BCR10S) Immediately Following Exercise at Weeks 4, 8, 12 and 16/Early Withdrawal
Description: The BCR10S score was collected immediately following completion of the 6-minute walk test. Baseline data was calculated as the average of the two BCR10S values obtained following the two 6MWD tests used in determining the Baseline 6MWD. If only one measurement was available, that measurement has been used. BCR10S scores ranges from 0 to 10 (0=nothing at all, 10=extremely strong). If participant's perception or feeling was stronger than "10", i.e "extremely strong", "Maximal" - a larger number could be used, e.g. 12 or still higher i.e "Absolute maximum"). Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: Baseline (Week 0); Weeks 4, 8, 12 and 16/Early Withdrawal
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Scores on a scale
  Week 4, n=15, 17 | 0.00 [-1.00 to 0.75] | -0.40 [-0.50 to 0.00]
  Week 8, n=14, 16 | 0.25 [-0.50 to 1.00] | -0.20 [-1.13 to 1.00]
  Week 12, n=13, 15 | 0.00 [-0.50 to 2.25] | -0.40 [-1.00 to 1.00]
  Week 16, n=13, 15 | 1.00 [-0.50 to 2.50] | -0.50 [-1.50 to 1.00]
  Early Withdrawal, n=3, 2 | 2.00 [-1.50 to 4.00] | -0.25 [-0.50 to 0.00]

5. Secondary Outcome: Number of Participants With Clinical Worsening of Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Description: Clinical worsening of CTEPH is defined by the time from randomization to the first occurrence of death, lung transplantation, hospitalization for CTEPH, atrial septostomy, addition of parenteral prostanoids, or study withdrawal due to two or more early escape criteria included: a decrease from Baseline of at least 20 percent in the distance walked during the six-minute walk test; an increase of one or more WHO functional class; worsening right ventricular failure (e.g., as indicated by increased jugular venous pressure; new/worsening hepatomegaly, ascites, or peripheral edema; worsening echocardiographic parameters such as tricuspid annulus plane systolic excursion (TAPSE) and Tissue Doppler Imaging of the tricuspid annulus); rapidly progressing cardiogenic, hepatic, or renal failure; refractory systolic hypotension (systolic blood pressure less than 85 millimeter of mercury [mmHg]).
Time Frame: From randomization to Week 16/Follow up visit (21 weeks)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Participants | 0 | 0

6. Secondary Outcome: Change From Baseline in Mean Right Atrial Pressure (mRAP) and Mean Pulmonary Artery Pressure (mPAP) at Week 16
Description: mPAP and mRAP are measures of cardiopulmonary hemodynamics. Baseline is the last value recorded on or prior to start of study treatment. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: Baseline (Week 0) and Week 16
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Millimeter of mercury (mmHg)
  mRAP, Week 16, n=11, 13 | -2.0 [-5.0 to 4.0] | -1.0 [-4.0 to 3.0]
  mPAP, Week 16, n=11, 12 | -6.0 [-10.0 to -1.0] | -3.0 [-11.6 to 2.0]

7. Secondary Outcome: Change From Baseline in Cardiac Index at Week 16
Description: Cardiac index is measure of cardiopulmonary hemodynamics. Baseline is the last value recorded on or prior to start of study treatment. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: Baseline (Week 0) and Week 16
Population: Intent-to-Treat (ITT) Population: comprised of all randomized participants who received at least 1 dose of study drug. Only those participants with available data at Baseline and the specified timepoint were summarized.
Measure: Median (Inter-Quartile Range); unit: Litre per minute per meter squared
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 11 | 12
Litre per minute per meter squared | 0.100 [-0.040 to 0.370] | 0.440 [0.030 to 1.015]

8. Secondary Outcome: Percent Change From Baseline in Plasma N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP)
Description: The ratio to baseline [BL] in NT-proBNP was calculated as the ratio of the value at the specified time-point to the BL value and was expressed as a percent change from BL. For each treatment group, the mean change from BL at the specified time-point was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the value at the specified time-point to BL on the original scale. The GM was expressed as a percentage (100*[GM - 1]). Standard Deviation(SD) is the SD of the mean change from baseline values on the log scale.
Time Frame: Baseline (Week 0); Weeks 4, 8, 12 and 16/Early Withdrawal
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Percent change
  Week 4, n=13, 15 | 43.6 (0.41) [12.0 to 84.1] | -15.8 (0.36) [-30.9 to 2.5]
  Week 8, n=13, 15 | 12.4 (0.49) [-16.2 to 50.8] | -23.3 (0.59) [-44.7 to 6.5]
  Week 12, n=12, 14 | 12.4 (0.59) [-22.9 to 63.9] | -21.9 (0.61) [-45.2 to 11.1]
  Week 16, n=12, 14 | 14.1 (0.55) [-19.5 to 61.6] | -29.4 (0.50) [-47.2 to -5.5]
  Early withdrawal, n=3, 2 | 35.7 (0.69) [-75.8 to 659.8] | -14.9 (0.31) [-95.0 to 1337.1]

9. Secondary Outcome: Change From Baseline in Quality of Life as Measured by Short Form 36 Health Survey (SF-36)
Description: The SF-36 v2 is a self-administered, health-related quality of life (QoL) metric. It is a 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health as well as 2 summary measures (Physical Health and Mental Health). Each domain is scored from 0 (poorer health) to 100 (better health). Change from Baseline was calculated as the post-Baseline score minus the Baseline score. The SF-36 data were collected, but after the study was terminated, not all endpoints listed in the protocol were analyzed, including the SF-36. This decision was documented in the reporting and analysis plan prior to database lock.
Time Frame: Baseline and up to Week 16/Early Withdrawal
Population: ITT Population
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect or important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Time Frame: From the start of study treatment and until follow up (Week 16/Follow up)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Participants
  Any AE | 15 | 11
  Any SAE | 1 | 0

11. Secondary Outcome: Change From Baseline in Haemoglobin Levels at Weeks 4, 8, 12, and 16/Early Withdrawal
Description: Haemoglobin levels were assessed at Screening, Baseline, Weeks 4, 8, 12, and 16/Early Withdrawal. Baseline is the last value recorded on or prior to start of study treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0); Weeks 4, 8, 12, and 16/Early Withdrawal
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Grams per liter
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Grams per liter
  Week 4, n=15, 15 | -2.0 [-5.0 to 6.0] | -5.0 [-10.0 to 2.0]
  Week 8, n=13, 16 | 0.0 [-8.0 to 3.0] | -7.5 [-10.5 to 1.5]
  Week 12, n=13, 14 | 2.0 [-6.0 to 8.0] | -5.0 [-9.0 to -1.0]
  Week 16, n=13, 15 | -3.0 [-10.0 to 2.0] | -6.0 [-9.0 to -3.0]
  Early withdrawal, n=3, 2 | -2.0 [-2.0 to 26.0] | -14.5 [-16.0 to -13.0]

12. Secondary Outcome: Change From Baseline in Haematocrit Levels at Weeks 4, 8, 12, and 16/Early Withdrawal
Description: Haematocrit levels were assessed at Screening, Baseline, Weeks 4, 8, 12, and 16/Early Withdrawal. Baseline is the last value recorded on or prior to start of study treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0); Weeks 4, 8, 12, and 16/Early Withdrawal
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Proportion of 1
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Proportion of 1
  Week 4, n=15, 15 | 0.000 [-0.016 to 0.015] | -0.015 [-0.033 to 0.012]
  Week 8, n=13, 16 | -0.003 [-0.026 to 0.014] | -0.021 [-0.035 to 0.003]
  Week 12, n=13, 14 | 0.007 [-0.017 to 0.022] | -0.023 [-0.029 to -0.004]
  Week 16, n=13, 15 | -0.007 [-0.031 to 0.004] | -0.019 [-0.033 to -0.003]
  Early withdrawal, n=3, 2 | -0.008 [-0.010 to 0.083] | -0.030 [-0.032 to -0.028]

13. Secondary Outcome: Number of Participants With Significant Liver Events at Weeks 4, 8, 12, and 16/Early Withdrawal
Description: A significant liver chemistry result is defined as any result which met the stopping criteria defined in the study protocol. Liver events were assessed at Screening, Baseline, Weeks 4, 8, 12, and 16/Early Withdrawal. Number of participants who reported a significant liver chemistry result are presented.
Time Frame: Weeks 4, 8, 12, and 16/Early Withdrawal
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Participants | 0 | 0

14. Secondary Outcome: Change From Baseline in Supine Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Assessed at Weeks 4, 8, 12, and 16/Early Withdrawal
Description: Vital sign measurements including supine systolic and diastolic blood pressure at Weeks 4, 8, 12, and 16/Early Withdrawal weeks. Supine blood pressure measurement was taken in a supine position having rested in this position for at least 10 minutes before each reading. Baseline is the last value recorded on or prior to start of study treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0); Weeks 4, 8, 12, and 16/Early Withdrawal
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
millimeter of mercury (mmHg)
  DBP, Week 4, n=15, 17 | 0.0 [-5.0 to 9.0] | -1.0 [-12.0 to 1.0]
  DBP, Week 8, n=14, 16 | 1.5 [-7.0 to 13.0] | -9.0 [-16.0 to -5.5]
  DBP, Week 12, n=13, 15 | 1.0 [0.0 to 7.0] | -8.0 [-14.0 to 5.0]
  DBP, Week 16, n=13, 15 | -2.0 [-10.0 to 8.0] | -10.0 [-16.0 to 3.0]
  DBP, Early Withdrawal, n=3, 2 | 16.0 [8.0 to 26.0] | -17.0 [-19.0 to -15.0]
  SBP, Week 4, n=15, 17 | 0.0 [-10.0 to 4.0] | -4.0 [-9.0 to 19.0]
  SBP, Week 8, n=14, 16 | 5.5 [-8.0 to 14.0] | -10.0 [-18.5 to -2.5]
  SBP, Week 12, n=13, 15 | -2.0 [-12.0 to 11.0] | -5.0 [-10.0 to 0.0]
  SBP, Week 16, n=13, 15 | -4.0 [-11.0 to 15.0] | -6.0 [-8.0 to 10.0]
  SBP, Early Withdrawal, n=3, 2 | 15.0 [10.0 to 18.0] | -8.0 [-16.0 to 0.0]

15. Secondary Outcome: Change From Baseline in Heart Rate Assessed at Weeks 4, 8, 12, and 16/Early Withdrawal
Description: Vital sign measurements including heart rate at Weeks 4, 8, 12, and 16/Early Withdrawal weeks. Baseline is the last value recorded on or prior to start of study treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0); Weeks 4, 8, 12, and 16/Early Withdrawal
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
beats per minute
  Week 4, n=15, 17 | 0.0 [-14.0 to 3.0] | 4.0 [-3.0 to 10.0]
  Week 8, n=14, 16 | -8.0 [-17.0 to 3.0] | 1.0 [-12.5 to 8.5]
  Week 12, n=13, 15 | -2.0 [-15.0 to 3.0] | 0.0 [-6.0 to 5.0]
  Week 16, n=13, 15 | 0.0 [-17.0 to 8.0] | -1.0 [-14.0 to 2.0]
  Early withdrawal, n=3, 2 | -6.0 [-24.0 to -3.0] | -18.0 [-32.0 to -4.0]

16. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters of Potential Clinical Concern Any Time Post Baseline
Description: Clinical chemistry parameters including alanine amino transferase (ALT), aspartate amino transferase (AST), creatinine, gamma glutamyl transferase (GGT) and total bilirubin (TB) assessed any time post Baseline. ALT: lower concern value and high concern value was considered as none and >=3xupper limit of normal (ULN) respectively. AST: lower concern value and high concern value was considered as none or >=3xULN respectively. creatinine: lower concern value and high concern value was considered as none and >=176.8 micromoles per liter (umol/L) respectively. GGT: lower concern value and high concern value was considered as none and >=3xULN respectively. For TB: lower concern value was none and high concern value was >=2xULN. Participants with both normal and low values were counted once under their worst case (Low). Participants with both normal and high values were counted once under their worst case (High). Participants with both high and low values are counted under both categories.
Time Frame: Baseline (Week 0), Weeks 4, 8, 12 and 16/early withdrawal,
Population: ITT Population
Measure: Number; unit: Participants
Groups:
- Placebo: Participants received a matching placebo tablet once daily for a period of 16 weeks.c
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Participants
  ALT, >clinical concern high | 0 | 0
  ALT, <clinical concern low | 0 | 0
  AST, >clinical concern high | 0 | 0
  AST, <clinical concern low | 0 | 0
  Creatinine, >clinical concern high | 0 | 0
  Creatinine, <clinical concern low | 0 | 0
  GGT, >clinical concern high | 1 | 1
  GGT, <clinical concern low | 0 | 0
  TB, >clinical concern high | 0 | 0
  TB, <clinical concern low | 0 | 0

17. Secondary Outcome: Number of Participants With Hematology Parameters of Potential Clinical Concern Any Time Post Baseline
Description: Hematology parameters including hemoglobin, international normalized ratio (INR), and platelet count assessed any time post Baseline. Baseline is the last value recorded on or prior to start of study treatment. For hemoglobin: lower concern value and high concern value was considered as <100 gram per liter (G/L) and none respectively. For INR: lower concern value and high concern value was considered as none or >5 prothrombin time respectively. For platelet count: lower concern value and high concern value was considered as <50 giga cells per liter (GI/L) and >500 GI/L respectively. Participants with both normal and low values were counted once under their worst case (Low). Participants with both normal and high values were counted once under their worst case (High). Participants with both high and low values are counted under both categories.
Time Frame: Baseline (Week 0), Weeks 4, 8, 12 and 16/early withdrawal
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 16 | 17
Participants
  Hemoglobin, >clinical concern high, n=16, 17 | 0 | 0
  Hemoglobin, <clinical concern low, n=16, 17 | 0 | 0
  INR, >clinical concern high, n=2, 0 | 0 | 0
  INR, <clinical concern low, n=2, 0 | 0 | 0
  Platelet count, >clinical concern high, n=16, 17 | 0 | 0
  Platelet count, <clinical concern low, n=16, 17 | 0 | 0

18. Secondary Outcome: Number of Participants With Testicular Function (Males Only) of Potential Clinical Concern Any Time Post Baseline
Description: For male participants testicular function (total testosterone, sex hormone binding globulin [SHBG-calculated free testosterone), follicle stimulating hormone (FSH), luteinizing hormone (LH), and inhibin B were assessed at Weeks 4 and 16/early withdrawal. The testicular function data were collected, but after the study was terminated, not all endpoints listed in the protocol were analyzed, including Testicular Function. This decision was documented in the reporting and analysis plan prior to database lock.
Time Frame: Baseline, Weeks 4 and 16/early withdrawal
Population: ITT Population
Arm/Group | Placebo | Ambrisentan 5mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment and until the follow up contact (Week 21)
Description: AEs and SAEs were collected from the members of ITT population which comprised of all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Ambrisentan 5mg
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/17
Other Adverse Events (participants affected / at risk) | 15/16 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Ambrisentan 5mg (N=17)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Ambrisentan 5mg (N=17)
Oedema peripheral (General disorders) | 2 | 3
Feeling abnormal (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Weight increased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.